CLINICAL TRIAL: NCT05488717
Title: The Effect of Art-Based Mandala on Mental Health in Bone Marrow Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysenur Uceriz (Other)
Collaborators: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Sponsor-Investigator, Aysenur Uceriz, Principal investigator, Istanbul University
Organization: Istanbul University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Master's thesis; Interventional research (Other: Istanbul Sabahattin Zaim University)
Record Dates: First submitted 2022-03-01; First posted 2022-08-04 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Mental Health; Bone Marrow Cancer; ART
MeSH Terms: conditions — Psychological Well-Being; Bone Marrow Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application (Experimental): Patients who are routinely scheduled for bone marrow transplantation are admitted to the unit one week before the transplant and treatment is started and transplantation is performed a week later. All patients in the intervention and control group will be filled out forms upon hospitalization after receiving their informed consent at the beginning of the study. Subsequently, patients in the intervention group will be given art-based mandala painting, which is sampled below, for 30 minutes for a week, accompanied by instrumental music featuring natural sounds in a room with light-heat control. Mandala painting templates and crayons will be provided by the researcher. The researcher will not intervene in any way other than time management during the preparation and painting of the environment. The researcher participated in training on art-based mandala and made preliminary preparations.
  No intervention will be made to the control group except for routine clinical applications.
  Interventions: Other: art-based mandala application

INTERVENTIONS:
Other: art-based mandala application — Patients who are routinely scheduled for bone marrow transplantation are admitted to the unit one week before the transplant and treatment is started and transplantation is performed a week later. All patients in the intervention and control group will be filled out forms upon hospitalization after receiving their informed consent at the beginning of the study. Subsequently, patients in the intervention group will be given art-based mandala painting, which is sampled below, for 30 minutes for a week, accompanied by instrumental music featuring natural sounds in a room with light-heat control. Mandala painting templates and crayons will be provided by the researcher. The researcher will not intervene in any way other than time management during the preparation and painting of the environment. The researcher participated in training on art-based mandala and made preliminary preparations.
  No intervention will be made to the control group except for routine clinical applications.

SUMMARY:
According to the World Health Organization (WHO), health is not only a state of complete well-being in terms of illness and disability, but also physical mental and social well-being. Mental health, on the other hand, is a state of goodness in which the individual is aware of his own abilities, copes with the normal tensions of life, can work productively and efficiently and contributes to the society in which he lives.

It has been shown in many studies that mental health problems negatively affect the existing disease process. For example, research shows an association between depression and anxiety and cardiovascular and cerebrovascular diseases . In the New York Health Survey, 10,000 individuals representing 33 communities were surveyed by phone; it was found that the general health status of people who reported significant emotional distress was three times worse than those who did not report it .

Realizing that mental health is more than just a disease will guide individuals and caregivers. Developing a more comprehensive clinical approach by focusing on a person's healthy, strengths, abilities and personal efforts is important in strengthening mental health. Applications for strengthening mental health include improving nutrition and housing conditions, increasing access to education, strengthening social networks, creating support environments.

In the acceptance and stability therapy study of Bash and Dirik with cancer, it was determined that the negative psychological symptoms of the patients decreased and their expectations of life and quality of life increased. In another study , it was determined that the spiritual support practices provided to 150 individuals with breast cancer positively affected the state of spiritual, psychological and physical well-being.

Cancer is a life-threatening disease that is common all over the world and affects the individual both physically and psychologically. Hematologic cancers are caused by bone marrow, the place of production of blood, and include diseases such as acute-chronic leukemias and multiple myelomas. Chemotherapy, radiotherapy, surgical methods in the treatment of hematologic cancers; hormonal and biological treatment and bone marrow transplantation (CIS) may be preferred.

Among the applications aimed at strengthening mental health are art-based applications (music therapy, applications for visual arts-painting, painting, mandala, clay works, etc.), collage, carving, sculpture, poetry therapy, etc.) as subheadings for the creation of supportive environments. we come across it. When the literature is examined, it is stated that the participation of individuals with art-based applications increases the adaptation process, helps them to find the meaning of life, increases their awareness of cancer and their life, is better adapted to disease and treatment, their emotional expression is more effective, and the state of spiritual and psychological well-being improves positively . Art-based applications provide a significant reduction in anxiety levels in adult cancer patients ; health-related quality of life . In other studies with cancer patients, it was found that art therapy practices reduce the feeling of anxiety and depression and cause a significant increase in health-related quality of life, patients feel more valued and strong, self-esteem increases, interpersonal relationships develop and they are more social .

DETAILED DESCRIPTION:
There is a limited number of studies, it is emphasized that art-based applications should be used as a complementary medicine method in cancer patients, nurses who have the most contact with patients in the care dimension use art-based applications to diagnose and control the symptoms. The aim of this study is to investigate the effect of art-based mandala on mental health in CIS patients who are cancer patient groups.

The research will be carried out at Istanbul University Istanbul Faculty of Medicine Department of Internal Medicine, Hematology Department Bone Marrow Service and Autologous Transplantation Unit.

Bone Marrow Service, which has a six-bed and isolated service feature, has 1 specialist doctor, 1 assistant doctor and 10 clinical nurses and an average of 18 allogenic bone marrow transplants are performed annually.

The twelve-bed Autologous Transplant Unit has 2 specialist doctors and 11 clinical nurses, and an average of 28 autologous transplants occur annually. Post-discharge complications are also monitored in the unit, which is not isolated service.

The study will be conducted between 15 January 2022 and 31 December 2022. The G*Power 3.1 program was used for power analysis calculations of the experimentally designed study. Taking into account Dogan's work, which is similar to the purpose and design of the study; the experimental group's desperation pretest score average of 5.05 (±3.72) to determine the sample size; final test score average 2.59 (±1.9); α margin of error: 0.05 and 1- β (power): 0.80. In this way, the sample size was calculated as 42; however, taking into account factors such as not participating in the study, leaving the study, etc.; design effect:1.1 and the final sample size was determined as 46. 46 patients to be included in the study; It was randomized with the IBM SPSS v.21 package program.The data will be collected with Patient Information Form , External Thermometer , Spielberger Continuous Anxiety Inventory, Beck Desperation Scale and Diener Psychological Well-Being Scale.

who are routinely scheduled for bone marrow transplantation are admitted to the unit one week before the transplant and treatment is started and transplantation is performed a week later. All patients in the intervention and control group will be filled out forms upon hospitalization after receiving their informed consent at the beginning of the study. Subsequently, patients in the intervention group will be given art-based mandala painting, which is sampled below, for 30 minutes for a week, accompanied by instrumental music featuring natural sounds in a room with light-heat control. Mandala painting templates and crayons will be provided by the researcher. The researcher will not intervene in any way other than time management during the preparation and painting of the environment. The researcher participated in training on art-based mandala and made preliminary preparations.

No intervention will be made to the control group except for routine clinical applications.

analysis of quantitative data obtained from the research will be done using IBM SPSS v.21 package program. For descriptive statistics for variables, mean, standard deviation, number (n) percentage (%) representation, and square-square test will be used for relationships between categorical variables. All analyses will be evaluated in a 95% reliability range. P<0.05 criteria will be taken for meaningfulness in all statistical analyses.

If the evaluation of both the experiment and the control group in the first interview, the comparison of evaluation scores before and after transplantation is provided with the assumption of normality, single-factor repetitive measurements are paired ANOVA test; if the assumption of normality is not provided, it will be examined by the Friedman test.

Permission will be obtained from the Scientific Research and Publication Ethics Board of Sabahttin Zaim University in Istanbul in order to carry out the research. The necessary permission will be obtained from the Department of Hematology of istanbul University Istanbul Faculty of Medicine, Department of Internal Medicine, where the research will be carried out. Those who are willing to participate in the study will be informed before the study and written consent will be obtained from the individuals. Since personal data will be collected in the research, all necessary measures will be taken to protect personal data in accordance with the Personal Data Protection Law No. 6698 and related legislation, and all necessary obligations will be carefully fulfilled.

ELIGIBILITY:
İnclusion criteria

* Being between the ages of 18 and 65
* Being in hospital for bone marrow transplantation
* Not having received any psychiatric diagnosis
* No physical barrier to painting mandala
* Being literate enough to fill the scales
* Having agreed to participate in the study

Exclusion criteria

* not be between the ages of 18-65
* Not being hospitalized for the bone marrow transplant process
* Having any psychiatric diagnosis
* Having a physical disability to paint mandalas
* Not being literate enough to fill in the scales
* to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Distress Thermometer | through study completion, an average of 1 year
  stress
  It is a visual analog scale in the form of a thermometer with numbers from 0 to 10. The scale is a 3-level thermometer scoring 0-10, and the patient is asked to indicate how much pressure they have felt during the past week; A score of 4 or above indicates that the patient has clinically significant distress.
State/ Trait Anxiety Inventory-STAI | through study completion, an average of 1 year
  trait anxiety
  7 of the trait anxiety statements (1, 6, 7, 10, 13, 16, 19) were correct, 13 (2, 3, 4, 5, 8, 9, 11, 12, 14, 15, 17, 18) , 20) is the opposite expression. While the reverse expressions expressing positive emotions are scored, those with a weight of 1 are converted to 4, and those with a weight of 4 are converted to 1. In direct statements expressing negative emotions, responses with a value of 4 indicate the height of anxiety. In the evaluation, the total score of the negative statements is subtracted from the total score of the positive statements, and a constant number of 35 is added to the value found. The resulting score; A score of 0-19 is considered no anxiety, a score of 20-39 is mild anxiety, 40-59 is moderate anxiety, 60-79 is severe anxiety, and a score of 80 and above is considered panic and crisis.
Beck Hopelessness Scale | through study completion, an average of 1 year
  Hopelessness
  The scale used to evaluate the hope and hopelessness status of the individual includes 20 statements with yes and no response options. The answer given to 11 items in the scale was yes (2, 4, 7, 9, 11, 12, 14, 16, 17, 18, 20. statements), and the answer to 9 items was no (1, 3, 5, 6, 8, 10, 13, 15, 19. phrases) are expected. A score of 1 is given if an expected response is given to each statement, and 0 is given if an unexpected response is given. The total score of the scale, ranging from 0 to 20, is determined by summing up the answers; A low score indicates a high level of hope, conversely, a high score indicates a low level of hope.
Psychological Well-Being Scale (PIOS) | through study completion, an average of 1 year
  psychological well-being
  All items in the scale are expressed positively; Each item is answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). The score obtained ranges from 8 (strongly disagree to all items) to 56 (strongly agree to all items). A high score indicates that the person has many psychological resources and strength, in other words, the level of psychological well-being is high.

SECONDARY OUTCOMES:
patient information form | through study completion, an average of 1 year
  It is a questionnaire consisting of 11 questions prepared by the researcher, including sociodemographic and medical information.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes